CLINICAL TRIAL: NCT02091661
Title: Radical Retropubic Prostatectomy Versus Conventional External Beam Radiotherapy for Clinically Localized Prostate Cancer
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: accrual too slow
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Savino M. Di Stasi, Associate Professor of Urology, University of Rome Tor Vergata
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UTV55/96
Record Dates: First submitted 2014-03-13; First posted 2014-03-19 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Prostate Cancer
Keywords: Clinically localized prostate cancer; Radical retropubic prostatectomy; External beam radiotherapy; Efficacy; Quality of life; adverse events
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radical retropubic prostatectomy (Active Comparator): The surgery arm underwent radical retropubic prostatectomy, performed by a technique described by Walsh.surgery started with dissection of the pelvic lymph nodes. If there were no signs of metastasis in frozen sections, the operation was continued with retropubic radical prostatectomy. The prostatectomy is performed in retrograde way, preserving the neurovascular bundles if feasible. The degree to which the surgeon preserve the nerves is categorized as non-nerve-sparing, unilateral nerve-sparing, or bilateral nerve-sparing.The operative time is about 2 to 3 hours and required hospital stay. The patient has a urinary catheter placed for 6 to 9 days to facilitate bladder emptying.
  Interventions: Procedure: Radical retropubic prostatectomy
- External beam radiotherapy (Active Comparator): External beam radiotherapy is carried out with intensity-modulated radiation technique. The treatment is designed to maximize the radiation dose to the prostate and seminal vesicles and minimize exposure to surrounding structures, including the bladder and rectum. Radiation to the prostate was delivered in fractionated doses divided over multiple treatments (180 to 200 centigray (cGy) daily fractions, 5 days per week) for a total dose to the prostate of 68 to 77 gray (Gy), prescribed at 90% to 100% of the isodose line.
  Interventions: Radiation: External beam radiotherapy

INTERVENTIONS:
Procedure: Radical retropubic prostatectomy — The surgery arm underwent radical retropubic prostatectomy, performed by a technique described by Walsh. The prostatectomy is performed in retrograde way, preserving the neurovascular bundles if feasible. The degree to which the surgeon preserve the nerves is categorized as non-nerve-sparing, unilateral nerve-sparing, or bilateral nerve-sparing. Pelvic lymph node dissection is performed if feasible. The operative time is about 2 to 3 hours and required hospital stay. The patient has a urinary catheter placed for 6 to 9 days to facilitate bladder emptying.
  Arms: Radical retropubic prostatectomy
Radiation: External beam radiotherapy — External beam radiotherapy is carried out with intensity-modulated radiation technique. The treatment is designed to maximize the radiation dose to the prostate and seminal vesicles and minimize exposure to surrounding structures, including the bladder and rectum. Radiation to the prostate was delivered in fractionated doses divided over multiple treatments (180 to 200 centigray (cGy) daily fractions, 5 days per week) for a total dose to the prostate of 68 to 77 gray (Gy), prescribed at 90% to 100% of the isodose line.
  Arms: External beam radiotherapy

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the two most established primary treatments for patients with clinically localized prostate cancer: radical retropubic prostatectomy, and external-beam radiotherapy. The primary aim is assessing biochemical disease-free survival, overall survival, and prostate cancer-specific survival. As secondary objectives quality of Life impact of treatments' side effects will be also assessed.

DETAILED DESCRIPTION:
Eligible patients had clinically localized (clinical TNM classification T1 or T2), biopsy-proven adenocarcinoma of the prostate and were randomly treated with RRP or EBRT. Exclusion criteria included prior treatment for prostate cancer, the presence of metastatic disease on imaging studies, the receipt of neoadjuvant androgen ablation before registration, and an inability to read or understand Italian language. The institutional review boards of every participating centre approved the study design. Every patient enrolled signed an informed-consent form approved by the institutional review boards. Clinical information collected from the medical record included pre-treatment serum prostate-specific antigen (PSA) level, clinical T classification, and biopsy Gleason score. Follow-up assessments were completed before treatment and every 3 months after treatment. Subjects who sought primary treatment elsewhere or did not return follow-up questionnaires beyond the initial assessment were excluded from this analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age 75 years or younger
* Diagnosis of prostate cancer, as verified by cytologic or histologic examination the tumor is well differentiated to moderately well differentiated
* Untreated, clinically localized prostate cancer, with a tumor stage of T1, or T2
* Prostate specific antigen (PSA) level of ≤10 ng/ml
* Bone scan with no abnormalities
* Health status that would permit radical prostatectomy
* Life expectancy of more than 10 years.

Exclusion Criteria:

* PSA >10 ng/ml
* Bone scan consistent with metastatic disease
* Other evidence that cancer of the prostate is not clinically localized
* Life expectancy less than 10 years
* Serum creatinine greater than 3 mg/dl
* Myocardial infarction within last 6 months
* Unstable angina Class III or IV
* Severe pulmonary disease
* Liver failure
* Severe dementia
* Debilitating illness Malignancies, except for nonmelanomatous skin cancer, in the last 5 years.

Max Age: 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 1997-01; Primary Completion 2001-09 (Actual); Study Completion 2020-03-24 (Estimated)

PRIMARY OUTCOMES:
Biochemical disease-free survival | up to 12 months
  Number of participants who are free of biochemical relapse after a specified duration of time. Biochemical recurrence is measured by PSA levels. The definition of biochemical recurrence was based on a review of the literature and consideration of clinical practice in the year 1997. Biochemical recurrence among patients who underwent radical prostatectomy (RP) was defined as a measurable serum PSA concentration 0.2 ng/ml or greater. The American Society for Therapeutic Radiology and Oncology (ASTRO) criteria were used to define progression after radiation therapy. The ASTRO consensus definition specifies progression as 3 consecutive increases in serum PSA documented at intervals of 6 or more months.

SECONDARY OUTCOMES:
•Perceived general health measured by the Medical Outcomes Study 36-Item Short Form (SF-36). | 1, 3, 6, 12 and 24 months after treatment.
  The Medical Outcomes Study 36-Item Short Form (SF-36) version 2 contains 36 items covering eight dimensions: physical functioning, role limitations due to physical health problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems and mental health. For each dimension, a score ranges from 0-100 (higher score indicate better health).Physical and mental component summaries are constructed, using recommended scoring algorithms. Summary scores are standardized to have a mean of 50 and standard deviation of 10 in the general population.
•Cancer specific Quality of Life measured by the Functional Assessment of Cancer Therapy - General and Prostate specific - (FACT-G and FACT-P, respectively). | 1, 3, 6, 12 and 24 months after treatment.
  The Functional Assessment of Cancer Therapy - General (FACT-G) version 4.0 was designed to measure Quality of Life in cancer patients. It consists of 27 items in 4 dimensions measuring Physical, Social/familial, Emotional, and Functional well-being. The Prostate module (FACT-P) is specific for patients with prostate cancer and contains 12 questions about urinary symptoms, and bowel and sexual function. Scores range from 0 to 108 on the FACT-G, and from 0 to 48 on the FACT-P, with 0 representing perfect health.
•Urinary symptoms measured by the International Prostate Symptom Score (IPSS). | 1, 3, 6, 12 and 24 months after treatment.
  The International Prostate Symptom Score (IPSS) was developed to assess the severity of lower urinary tract symptoms associated to Benign Prostatic Hyperplasia and has also been applied to other conditions that cause lower urinary tract symptoms (LUTS). The IPSS consists of a total of seven questions that deal with voiding symptoms (incomplete empty, intermittency, weak stream and straining to void) and storage symptoms (frequency, urgency and nocturia) and an additional question to measure quality of life. The score ranges from 0 to 35, with lower scores denoting a better health state.
•Sexual symptoms measured by the International Index of Erectile Function (IIES). | 1, 3, 6, 12 and 24 months after treatment.
  The International Index of Erectile Function (IIES) is a 15-item, self-administered questionnaire scale for the assessment of erectile function. Scores range from 5 to 75, with higher scores denoting a better sexual function.
Overall survival. | 5, 7 and 10 years after treatment and every 5 years thereafter.
  Number of participants who are alive after a specified duration of time.
Prostate cancer-specific survival | 3, 5, and 10 years after treatment and then every 5 years thereafter
  Number of participants who are not dead due to prostate cancer after a specified duration of time

CONTACTS AND LOCATIONS:
Overall Officials: Savino M. Di Stasi, MD, PhD, Study Chair — Tor Vergata University of Rome